CLINICAL TRIAL: NCT02325297
Title: "Impacts of the Letter of Condolence to the Bereaved Families Experience After a Death in ICU " - Study Famirea 22
Acronym: Famirea 22
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Famirea22
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Death; Mourning
Keywords: Intensive care unit
MeSH Terms: conditions — Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Letter of condolence (Experimental): Letter of condolence 15 days after the death of the relative.
  Interventions: Other: Letter of condolence
- No letter of condolence (No Intervention): No letter of condolence

INTERVENTIONS:
Other: Letter of condolence
  Arms: Letter of condolence

SUMMARY:
After the death of a patient in the hyper-technical context of intensive care, his relatives are particularly vulnerable and often exhibit symptoms of anxiety, depression, post traumatic stress and complicated grief. The first results of a qualitative study Famiréa current (CAESAR) support the idea that the bereaved relatives suffer from persistent misunderstandings and a feeling of abandonment of the resuscitation team. Many families suggest the need for contact with the team after the patient's death. The letter of condolence received by some families allowed them to feel recognized in their pain resuscitation teams. This has led us to ask the question of post-death monitoring and interest to send to bereaved relatives a letter of condolence, as recommended by the American consensus conference in 2004 on good palliative care. This strategy would allow the recognition of both close to the pain but also the strong bond that united the resuscitation team. The hypothesis of the study is that the post-death followed in the form of a letter of condolence sent by the intensive care physician who was in charge of the patient, could reduce the risk of having symptoms of anxiety / depression and post-traumatic stress and reduce the rate of complicated grief.

Famirea 22 is randomized clinical trial aimin to compare two bereaved groups: one group who did not receive a letter of condolence and a group that received a letter of condolence 15 days after the death.

ELIGIBILITY:
Inclusion Criteria:

* death of a relative patient in intensive care whose relatives were interviewed at least once by resuscitation team
* death of an adult relative patient
* ICU stay of the relative patient more than 2 days

Exclusion Criteria:

* death of a pregnant woman
* opposition to the use of its data by the patient
* relative does not speak French
* refusal of the relative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
HADS (Hospital Anxiety and Depression Scale) | 1 month

SECONDARY OUTCOMES:
Caesar scale | 1 month
  a questionnaire describing ICU end-of-life practices and satisfaction with the patient's care, communication, and symptom management during the dying process.
IES-R (Impact of Event Scale, Revised) | 6 months
ICG (Inventory of Complicated grief) | 6 months
HADS (Hospital Anxiety and Depression Scale) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Louis Hospital, Paris, Paris, France

REFERENCES:
- [Derived] Kentish-Barnes N, Chevret S, Champigneulle B, Thirion M, Souppart V, Gilbert M, Lesieur O, Renault A, Garrouste-Orgeas M, Argaud L, Venot M, Demoule A, Guisset O, Vinatier I, Troche G, Massot J, Jaber S, Bornstain C, Gaday V, Robert R, Rigaud JP, Cinotti R, Adda M, Thomas F, Calvet L, Galon M, Cohen-Solal Z, Cariou A, Azoulay E; Famirea Study Group. Effect of a condolence letter on grief symptoms among relatives of patients who died in the ICU: a randomized clinical trial. Intensive Care Med. 2017 Apr;43(4):473-484. doi: 10.1007/s00134-016-4669-9. Epub 2017 Feb 14. PMID 28197680
- [Derived] Kentish-Barnes N, Chevret S, Azoulay E. Impact of the condolence letter on the experience of bereaved families after a death in intensive care: study protocol for a randomized controlled trial. Trials. 2016 Feb 20;17(1):102. doi: 10.1186/s13063-016-1212-9. PMID 26897630